CLINICAL TRIAL: NCT01841736
Title: Prospective Randomized Phase II Trial of Pazopanib (NSC #737754) Versus Placebo in Patients With Progressive Carcinoid Tumors
Brief Title: Pazopanib Hydrochloride in Treating Patients With Progressive Carcinoid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00831; NCI-2013-00831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALLIANCE A021202; CALGB-A021202; A021202 (Other: Alliance for Clinical Trials in Oncology); A021202 (Other: CTEP); U10CA031946 (NIH); U10CA180821 (NIH); U10CA180830 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Foregut Neuroendocrine Tumor; Hindgut Neuroendocrine Tumor; Metastatic Digestive System Neuroendocrine Tumor G1; Metastatic Neuroendocrine Tumor; Midgut Neuroendocrine Tumor G1; Neuroendocrine Tumor G2; Recurrent Digestive System Neuroendocrine Tumor G1; Regional Digestive System Neuroendocrine Tumor G1
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; pazopanib; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening. Patients also undergo CT, MRI, and chest x-ray throughout the trial. Patients may optionally undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Pazopanib Hydrochloride; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. At the time of progressive disease, patients may cross-over to Arm I. Patients undergo ECHO or MUGA during screening. Patients also undergo CT, MRI, and chest x-ray throughout the trial. Patients may optionally undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Other: Placebo Administration; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW 786034B; GW-786034B; GW786034B; Pazopater; Votrient
  Arms: Arm I (pazopanib hydrochloride)
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This randomized phase II trial studies how well pazopanib hydrochloride works in treating patients with carcinoid tumors that are growing, spreading, or getting worse. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. For patients with progressive carcinoid tumors, progression-free survival (PFS defined by central review according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) will be compared between patients randomized to treatment with pazopanib (pazopanib hydrochloride) versus placebo.

SECONDARY OBJECTIVES:

I. Overall survival (OS) will be compared between treatment arms. II. Objective response rate, duration of response, and time to treatment failure will be compared between treatment arms.

III. Progression free survival (PFS) as assessed by central radiology review and local radiology review will be compared overall and within treatment arms.

IV. Safety and tolerability of treatment with pazopanib/placebo will be evaluated within each treatment arm.

V. PFS and other indicators of efficacy will be estimated in patients who crossover to pazopanib from placebo.

VI. To determine the turn-around time for timely adjudicated central review. VII. To characterize the nature of discordance between local and central radiology review in assessment of progression.

VIII. To characterize the type and rate of progression in carcinoid (at study entry, on-study, and at progression).

IX. To develop new methods for modeling carcinoid growth and detecting treatment effects, and to perform simulations that advance new clinical trial designs to apply to future trials of carcinoid therapeutics.

X. To assess for differences in quality of life (QOL)-related domains between the two treatment groups (pazopanib versus placebo).

XI. To determine if the more brief measures of QOL-related domains provide comparable information to that which is provided by the longer assessments (European Organization for Research and Treatment of Cancer [EORTC], neuroendocrine tumors [NET]21).

XII. To provide validation data for the EORTC NET21 module in terms of responsiveness over time and differences across arms.

XIII. To determine whether components of the plasma angiome panel that have been shown to be predictive previously (interleukin-6 [IL-6] and vascular endothelial growth factor [VEGF]-D) are predictive of a therapeutic advantage for pazopanib treatment in baseline samples from the patients treated on A021202.

XIV. To determine whether other components of the plasma angiome panel tested (not IL-6 and VEGF-D) are predictive of a therapeutic advantage for pazopanib treatment in baseline samples from the patients treated on A021202.

XV. To evaluate the changes in the plasma angiome markers after treatment with or without pazopanib over time.

EXPLORATORY OBJECTIVES:

I. PFS at 6 months will be estimated within each treatment arm. II. Biochemical response (for chromogranin A, defined as a decrease of 50% or more in chromogranin A levels from baseline and for 5-hydroxyindoleacetic acid [5-HIAA], defined as a decrease of 50% or more in urinary 5-HIAA levels from baseline) will be compared between treatment arms among patients with elevated baseline levels of chromogranin A (CGA) and 5-HIAA.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and chest x-ray throughout the trial. Patients may optionally undergo blood sample collection during screening and on study.

ARM II: Patients receive placebo PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. At the time of progressive disease, patients may cross-over to Arm I. Patients undergo ECHO or MUGA during screening. Patients also undergo CT, MRI, and chest x-ray throughout the trial. Patients may optionally undergo blood sample collection during screening and on study.

After completion of study treatment, patients are followed up every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Low- or intermediate-grade neuroendocrine carcinoma, including the following subtypes: carcinoid tumor, low- to intermediate-grade or well- to moderately-differentiated neuroendocrine carcinoma or tumor, atypical carcinoid tumor; documentation from a primary tumor or metastatic site is sufficient; patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid tumor, or goblet cell carcinoid tumor are not eligible
* Locally unresectable or metastatic carcinoid tumors
* Patients must have histologic documentation or clinical evidence of a carcinoid tumor of primary site (including foregut, midgut, hindgut or other non-pancreatic site); tumors of unknown primary site are eligible provided the treating physician does not suspect medullary thyroid cancer, pancreatic neuroendocrine tumor, paraganglioma, or pheochromocytoma; unknown primary tumors will be classified as small bowel tumors for the purpose of stratification; functional (associated with a clinical syndrome) or nonfunctional tumors are allowed; target lesions must have shown disease progression if therapy included peptide receptor radiotherapy (PRRT) and PRRT must be completed at least 8 weeks prior to registration
* Radiological evidence for progressive disease (measurable or non-measurable) within 12 months prior to registration; patients who have received anti-tumor therapy during the past 12 months (including octreotide analogs) must have had radiological documentation of progression of disease while on or after receiving therapy
* No known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage; patients with lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (computed tomography [CT] with contrast is strongly recommended to evaluate such lesions); patients with large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed
* Patients must have measurable disease per RECIST 1.1 by computed tomography (CT) scan or magnetic resonance imaging (MRI); lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as >= 1 cm with CT or MRI (or >= 1.5 cm for lymph nodes); index lesions for the purpose of RECIST 1.1 measurements will not be selected from within the radiation therapy treatment field; however, if there is evidence of disease progression within the radiation treatment field, measurement of the progressing lesions will be documented
* No prior treatment with an inhibitor of vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR)
* Prior treatment (somatostatin analogs excepted) must be completed at least 2 weeks prior to registration; in addition, prior treatment (somatostatin analogs excepted) must be completed at least 4 weeks prior to initiation of study drug; treatment-related toxicities must have improved to =< grade 1 prior to registration, with the exception of alopecia
* Concurrent use of somatostatin analogs (SSTa) is allowed, provided that the patient is on a stable dose for at least two months and progressive disease on somatostatin analog has been documented; progression on octreotide is required for patients with tumors arising in the midgut
* Prior treatment with embolization (including bland embolization, chemoembolization, and selective internal radiation therapy) or ablative therapies is allowed if measurable disease remains outside of the treated area or there is documented disease progression in a treated site; there is no limit on the prior number of procedures; prior liver-directed or other ablative treatment must be completed at least 8 weeks prior to registration; index lesions for the purpose of RECIST 1.1 measurements will not be selected from within the radiation therapy treatment field; however, if there is evidence of disease progression within the radiation treatment field, measurement of the progressing lesions will be documented
* Patients should have completed any major surgery >= 4 weeks prior to registration and must have completed any minor surgery >= 2 weeks prior to registration; patients must have fully recovered from the procedure

  * The following are examples of procedures considered to be minor: port placement, laparoscopy, thoracoscopy, bronchoscopy, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and dental extraction procedures
  * Insertion of a vascular access device, thoracentesis, paracentesis, and endoscopic ultrasonographic procedures are not considered to be major or minor surgeries
* No concurrent condition resulting in immune compromise, including chronic treatment with corticosteroids or other immunosuppressive agents
* No clinical evidence of central nervous system (CNS) metastases (including carcinomatous meningitis) at baseline, with the exception of those patients who have previously-treated CNS metastases (surgery +/- radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) had no requirement for steroids or enzyme-inducing anticonvulsants within 6 months prior to registration
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to registration
* No clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding within 28 days prior to registration including, but not limited to:

  * Active peptic ulcer
  * Known endoluminal metastatic lesion(s) with history of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
* No history of serious (i.e., requiring active medical therapy with medication or medical device under the supervision of a physician) non-healing wound, ulcer, trauma, or bone fracture within 28 days prior to study entry
* Patients with a history of hypertension must have blood pressure that is adequately controlled on antihypertensives; (< 140/90 mm Hg)
* No symptomatic congestive heart failure (New York Heart Association class II, III, or IV) within 6 months prior to registration
* No arterial thrombotic events within 6 months of registration, including transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral arterial thrombus, myocardial infarction (MI), or unstable angina or angina requiring surgical or medical intervention in 6 months prior to registration; patients with clinically significant peripheral artery disease (i.e., claudication on less than one block) are ineligible; patients who have experienced a deep venous thrombosis or pulmonary embolus within 6 months prior to registration must be on stable therapeutic anticoagulation for at least 6 weeks prior to enrollment of this study
* Patients on therapeutic anticoagulation with low molecular weight heparins, fondaparinux, rivaroxaban or warfarin are eligible, provided that they are on a stable dose of anticoagulants; patients who are currently receiving antiplatelet therapy of prasugrel or clopidogrel or antiaggregation agents (e.g., eptifibatide, epoprostenol, dipyridamole) or low doses of acetylsalicylic acid (up to 100 mg daily) are also eligible
* No ongoing cardiac dysrhythmias, atrial fibrillation, or prolongation of corrected QT (QTc) interval to > 480 msec
* No evidence of active bleeding, bleeding diathesis, or hemoptysis (>= 1/2 teaspoon of red blood) within 8 weeks prior to registration
* No currently unstable angina and/or uncontrolled cardiac arrhythmias
* Patients with symptomatic peripheral vascular disease are ineligible
* Ejection fraction on echocardiogram (Echo) or multi gated acquisition scan (MUGA) > 50%
* Chronic concomitant treatment with strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) is not allowed on this trial; patients on strong CYP3A4 inhibitors must discontinue the drug 14 days prior to the start of study treatment
* Women must not be pregnant or nursing; women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to registration; women of child-bearing potential include any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >= 12 consecutive months; or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL)
* Age >= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Granulocytes >= 1,500/mcL
* Platelets >= 100,000/mcL
* International normalized ratio (INR) =< 1.2 X upper limit of normal (ULN); only required for patients receiving anticoagulant therapy; patients are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* QTc =< 480 msecs
* Thyroid stimulating hormone (TSH) within normal limits (WNL); medications for thyroid dysfunction are allowed as long as TSH is normal at registration; in patients with abnormal TSH, if the free thyroxine (free T4) and free thyroxine index (FTI) are normal and patient is clinically euthyroid, patient is eligible
* Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) & alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN; concomitant elevations in bilirubin and AST/ALT above 1.0 X ULN are NOT permitted; also, if liver metastases are present, AST & ALT =< 5 x ULN is allowed
* Serum creatinine =< 1.5 x ULN
* Urine protein to creatinine ratio < 1, or, 24-hour urine protein < 1 g; if urine protein to creatinine (UPC) >= 1, then a 24-hour urine protein must be assessed; patients must have a 24-hour urine protein value < 1 g to be eligible; use of urine dipstick for renal function assessment is not acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2026-09-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Bergsland, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (424):
- United States (413):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Newman Regional Health, Emporia, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - University of Rochester, Rochester, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (11):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Vitalite Health Network - Dr Leon Richard Oncology Centre, Moncton, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Bergsland EK, Geyer S, Asmis TR, Behr SC, Kuebler JP, Kumthekar P, Mazza G, Maitland ML, Niedzwiecki D, Nixon AB, Schwartz LH, Strosberg JR, Venook AP, O'Reilly EM, Meyerhardt JA. Randomized Phase II Trial of Pazopanib Versus Placebo in Patients With Advanced Extrapancreatic Neuroendocrine Tumors (Alliance A021202). J Clin Oncol. 2025 Oct 10;43(29):3170-3183. doi: 10.1200/JCO-24-02644. Epub 2025 Sep 3. PMID 40902132

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Pazopanib Hydrochloride): Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo): Patients receive 800 mg placebo PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. At the time of progressive disease, patients may cross-over to Arm I.
Period: Overall Study
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Started | 97 | 74
Crossover (Crossed over for pazopanib following disease progression on placebo) | 0 | 49
Completed (Included in efficacy analysis) | 97 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 97 | 74 | 171
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 89] | 63 [37 to 85] | 63 [33 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 33 | 96
  Male | 34 | 41 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (White vs Non-White): Non-White | 20 | 12 | 32
  Race (White vs Non-White): White | 77 | 62 | 139
ECOG Performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 48 | 41 | 89
    1 | 48 | 33 | 81
    missing data | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS will be measured from date of patient entry until documented progression of disease as determined by central review or death from any cause. If a patient does not have a documented date of progression or death, then PFS will be censored at the date of last adequate assessment. PFS will be estimated within treatment arm using the Kaplan-Meier method. Progression is defined as any new lesion or increase by ≥20% of previously involved sites from nadir based on RECIST criteria.
Time Frame: From date of patient entry until documented progression of disease or death from any cause, assessed up to 5 years
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 97 | 74
months | 11.6 [11.0 to 13.0] | 8.5 [5.8 to 8.9]
Statistical Analysis 1: Comparison: Arm I (Pazopanib Hydrochloride) vs Arm II (Placebo); Test type: Superiority; p = 0.0005, Log Rank; Stratified log rank; Hazard Ratio (HR) = 0.53, 80% CI 2-sided [0.42 to 0.69]

2. Secondary Outcome: Best Response
Description: The best response per RECIST 1.1 criteria of participants receiving randomized treatment assignment. Complete response (CR): Disappearance of all evidence of disease, Partial response (PR): Regression of measurable disease and no new sites, Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum diameters while on study. Progressive disease (PD): Any new lesion or increase by ≥20% of previously involved sites from nadir. Note that those considered evaluable for best response here were those who had disease measurements while on treatment. Those who discontinued therapy early prior to a disease evaluation were not included.
Time Frame: Up to 5 years
Population: Per protocol, patients who crossover from placebo to active therapy at the time of progression will be followed for a second progression unless they withdraw from treatment for other reasons; in that case they will be followed for toxicity and survival only; thus response data are not available for "Placebo Crossover" group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 97 | 74
Participants
  Partial Response | 2 | 0
  Stable Disease | 70 | 54
  Progressive Disease | 4 | 14
  Not Evaluable | 21 | 6

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) will be measured from randomization until death from any cause. A patient who is alive at the time of the statistical analysis will be considered censored at the last date of known contact. OS will be estimated by the Kaplan-Meier method within each treatment arm.
Time Frame: From randomization until death from any cause, assessed up to 5 years
Population: This trial only has two arms ((Arm I (pazopanib hydrochloride) and Arm II (placebo)) that were analyzed. Pazopanib hydrochloride and Pazopanib are synonyms and Pazopanib was deleted. Per protocol, OS will be estimated by the Kaplan-Meier method within each treatment arm. OS for placebo patients who crossed over is not a specified outcome measure.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 97 | 74
months | 41.3 [31.9 to 44.8] | 42.4 [29.7 to 50.8]
Statistical Analysis 1: Comparison: Arm I (Pazopanib Hydrochloride) vs Arm II (Placebo); Test type: Superiority; p = 0.7, Log Rank; Stratified Log-Rank; Hazard Ratio (HR) = 1.13, 80% CI 2-sided [0.84 to 1.51]

4. Secondary Outcome: Duration of Response for the Subset of Patients With a Confirmed Complete Response or Partial Response
Description: Duration of response is defined as the time from documented response to time of progression and/or death. This time-to-event outcome will be summarized descriptively using the methods of Kaplan and Meier to characterize the cohort and distribution of this outcome.
Time Frame: From first documented evidence of complete response or partial response until first documented disease progression or death from any cause, assessed up to 5 years
Population: Duration of Response won't be a viable analysis as there aren't enough patients with partial responses
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 3 | 1
months | 11.9 [9.8 to NA] — There aren't enough patients with partial responses | 13.8 [NA to NA] — There aren't enough patients with partial responses

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from randomization to the time that treatment is terminated, including the reasons of disease progression, adverse events, withdrawal from study, or death. This time-to-event outcome will be evaluated using the methods of Kaplan and Meier.
Time Frame: From randomization until termination of protocol therapy for any reason including progression of disease, adverse events, and death, assessed up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 97 | 74
months | 8.5 [0.9 to 53.8] | 8.6 [0.3 to 48.0]

6. Other Pre Specified Outcome: Time to Second Progression for Patients Who Crossover From Placebo to Active Therapy
Description: Time to second progression will be defined as the progression free survival from crossover re-registration to documented progression of disease as determined by central review or death from any cause. If a patient does not have a documented date of progression or death, then PFS will be censored at the date of last adequate assessment. PFS will be estimated within treatment arm using the Kaplan-Meier method. Progression is defined as any new lesion or increase by ≥20% of previously involved sites from nadir based on RECIST criteria.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Placebo Crossover: Participants in Arm II (Placebo) who crossed over to receive pazopanib hydrochloride after having documented progression on Placebo.
Arm/Group | Placebo Crossover
Number analyzed (Participants) | 49
months | 12.1 [5.9 to 19.5]

7. Other Pre Specified Outcome: PFS Within Each Arm
Description: Kaplan-Meier methods will be used including calculations of 95% confidence intervals.
Time Frame: At 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Biochemical Response
Description: Biochemical response (for chromogranin A, defined as a decrease of 50% or more in chromogranin A levels from baseline, and for 5-hydroxyindoleacetic acid [5-HIAA], defined as a decrease of 50% or more in urinary 5-HIAA levels from baseline) will be compared between treatment arms among patients with elevated baseline levels of serum chromogranin A (CGA) and 5-HIAA.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo) | Placebo Crossover
All-Cause Mortality (participants affected / at risk) | 49/97 | 40/74 | 29/49
Serious Adverse Events (participants affected / at risk) | 16/97 | 3/74 | 2/49
Other Adverse Events (participants affected / at risk) | 90/97 | 71/74 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pazopanib Hydrochloride) (N=97) | Arm II (Placebo) (N=74) | Placebo Crossover (N=49)
Death NOS (General disorders) | 10 (10) | 2 (2) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pazopanib Hydrochloride) (N=97) | Arm II (Placebo) (N=74) | Placebo Crossover (N=49)
Anemia (Blood and lymphatic system disorders) | 17 (67) | 13 (90) | 12 (28)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 2 (7) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (5) | 2 (2) | 2 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (6) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (5) | 1 (11) | 2 (6)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (8) | 2 (11) | 2 (10)
Tricuspid valve disease (Cardiac disorders) | 2 (13) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 3 (5) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (38) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (10)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (22) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 5 (11) | 1 (1) | 1 (5)
Hypoparathyroidism (Endocrine disorders) | 1 (7) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 11 (55) | 2 (3) | 9 (13)
Blurred vision (Eye disorders) | 4 (5) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (4) | 0 (0) | 2 (3)
Floaters (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Night blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 1 (5) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (4) | 3 (9) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 23 (93) | 20 (35) | 13 (44)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 4 (12) | 3 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (14) | 8 (26) | 4 (11)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 65 (664) | 42 (308) | 35 (206)
Dry mouth (Gastrointestinal disorders) | 7 (41) | 0 (0) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (30) | 4 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (49) | 3 (4) | 3 (5)
Gastric hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (12) | 3 (5) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 9 (56) | 4 (4) | 2 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 10 (17) | 6 (12) | 5 (10)
Nausea (Gastrointestinal disorders) | 71 (326) | 37 (131) | 28 (107)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 (7) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 5 (7) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Visceral arterial ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 27 (53) | 10 (31) | 12 (21)
Chills (General disorders) | 4 (5) | 2 (2) | 3 (3)
Edema face (General disorders) | 2 (4) | 0 (0) | 1 (2)
Edema limbs (General disorders) | 12 (46) | 5 (28) | 9 (25)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 80 (786) | 58 (370) | 42 (292)
Fever (General disorders) | 3 (3) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 2 (3) | 3 (3) | 1 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 6 (10) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (14) | 2 (3) | 2 (2)
Pain (General disorders) | 7 (10) | 4 (25) | 8 (12)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (8) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (5) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (18) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 2 (2) | 4 (4)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 7 (29) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 4 (4) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 (7) | 0 (0) | 0 (0)
Urostomy obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 54 (167) | 25 (97) | 27 (130)
Alkaline phosphatase increased (Investigations) | 14 (29) | 14 (49) | 13 (51)
Aspartate aminotransferase increased (Investigations) | 61 (229) | 26 (102) | 28 (129)
Blood bilirubin increased (Investigations) | 28 (103) | 15 (58) | 18 (91)
Creatinine increased (Investigations) | 8 (14) | 6 (15) | 2 (3)
INR increased (Investigations) | 2 (6) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 3 (34) | 1 (1) | 2 (11)
Lipase increased (Investigations) | 3 (16) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (64) | 6 (46) | 6 (18)
Neutrophil count decreased (Investigations) | 30 (134) | 3 (5) | 12 (46)
Platelet count decreased (Investigations) | 21 (156) | 5 (12) | 9 (21)
Serum amylase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight loss (Investigations) | 18 (99) | 7 (8) | 8 (30)
White blood cell decreased (Investigations) | 21 (133) | 4 (23) | 6 (28)
Anorexia (Metabolism and nutrition disorders) | 24 (56) | 12 (30) | 14 (37)
Dehydration (Metabolism and nutrition disorders) | 8 (10) | 4 (4) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (63) | 12 (72) | 5 (23)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (32) | 6 (23) | 4 (16)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (4)
Hypernatremia (Metabolism and nutrition disorders) | 5 (9) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (70) | 5 (8) | 6 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (30) | 5 (13) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (10) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (19) | 4 (6) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (49) | 7 (30) | 4 (17)
Hyponatremia (Metabolism and nutrition disorders) | 8 (13) | 3 (3) | 6 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (12) | 4 (14) | 4 (19)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 2 (3) | 2 (13) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (31) | 2 (20) | 3 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (31) | 10 (32) | 6 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (16) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (16) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (20) | 5 (11) | 5 (12)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (13) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (13) | 4 (21) | 3 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (3)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (10) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (64) | 3 (6) | 5 (17)
Leukemia second to oncology chemo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (7) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 12 (23) | 6 (27) | 5 (15)
Dysgeusia (Nervous system disorders) | 14 (84) | 1 (1) | 2 (8)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 19 (47) | 7 (32) | 6 (17)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (16) | 1 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
Neuralgia (Nervous system disorders) | 1 (8) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (12) | 6 (8) | 1 (8)
Presyncope (Nervous system disorders) | 1 (1) | 1 (2) | 1 (4)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (22) | 1 (8)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 2 (4) | 2 (2) | 1 (2)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (15) | 3 (4)
Confusion (Psychiatric disorders) | 3 (3) | 1 (21) | 2 (9)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (13) | 2 (12) | 1 (7)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (35) | 8 (31) | 6 (25)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2) | 1 (3) | 1 (7)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 8 (27) | 4 (6) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (4) | 1 (1) | 2 (3)
Renal calculi (Renal and urinary disorders) | 1 (1) | 2 (4) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (28) | 1 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (9) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (8) | 1 (4)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (38) | 3 (4) | 4 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (54) | 3 (4) | 4 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (154) | 1 (1) | 2 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (13) | 4 (9) | 3 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (15) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 6 (27) | 1 (1) | 2 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (9) | 4 (11) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (26) | 1 (1) | 3 (17)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 21 (237) | 8 (31) | 8 (28)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (9) | 0 (0) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (34) | 0 (0) | 2 (24)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 4 (12) | 5 (23) | 5 (22)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 7 (25) | 5 (35) | 4 (15)
Hypertension (Vascular disorders) | 68 (695) | 46 (346) | 35 (215)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT01841736/Prot_SAP_000.pdf